CLINICAL TRIAL: NCT01756651
Title: A Prospective Study Comparing the Efficacy and Safety of 100 mcg and 200 mcg of Intranasal Fentanyl Pectin Spray as an Analgesic in Adult Males Undergoing Outpatient Cystoscopic Procedures
Brief Title: Intranasal Fentanyl for Management of Pain Associated With Cystoscopic Procedures
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Richard C Reznichek, MD (Other)
Collaborators: Depomed (Industry)
Responsible Party: Sponsor-Investigator, Richard C Reznichek, MD, Medical Doctor, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Organization: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20812-01
Record Dates: First submitted 2012-12-20; First posted 2012-12-27 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Other Acute Pain; Pain Experienced During Cystoscopy
Keywords: Intranasal fentanyl; Cystoscopy
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intranasal Fentanyl 100mcg (Experimental): fentanyl pectin nasal spray 100mcg
  Interventions: Drug: Fentanyl pectin
- Intranasal Fentanyl 200mcg (Experimental): fentanyl pectin nasal spray 200mcg
  Interventions: Drug: Fentanyl pectin

INTERVENTIONS:
Drug: Fentanyl pectin — comparison of Intranasal fentanyl 100mcg vs 200 mcg.
  Other Names: Lazanda; Fentanyl

SUMMARY:
The purpose of this study is to assess the safety and efficacy of intranasally-administrated fentanyl pectin spray (Lazanda®)given to decrease the pain during cystoscopy (the passage of a telescopic instrument into the bladder for purpose of diagnosing the cause of blood in the urine, urinary complaints or any other problems with the urinary bladder). The current standard practice is to use Lidocaine jelly (a local anesthetic) given through the urethra to lubricate and decrease local pain. In this study, an additional medicine (Lazanda®) is used to reduce pain that occurs during and after the above procedure.

DETAILED DESCRIPTION:
In this prospective study, twenty subjects will be enrolled. The first ten will receive a dose of 100mcg pectin fentanyl nasal spray (Lazanda®). The second ten will receive a dose of 200mcg pectin fentanyl nasal spray (Lazanda®) if the 100mcg was well tolerated in the first ten. In all cases, Lidocaine jelly is used as an local anesthetic in the urethra.

ELIGIBILITY:
Inclusion Criteria:

1. Male adult patients scheduled for cystoscopy; additional procedures (e.g. ureteral stent placement, stent exchange, bladder biopsy, retrograde pyelogram) may be included.

Exclusion Criteria:

1. History of analgesic abuse or opioid tolerance
2. Allergy to fentanyl or to any of the components of Lazanda®
3. Acute/chronic nasal problems such as rhinitis or sinusitis
4. Acute bronchial asthma / upper airway obstruction
5. Presence of bradycardia or history of seizures
6. Concomitant use of drugs that inhibit cytochrome P450 isoenzyme 3A4 (e.g., ritonavir, ketoconazole, itraconazole, troleandomycin, clarithromycin, nelfinavir, nefazodone, amprenavir, aprepitant, diltiazem, erythromycin, fluconazole, fosamprenavir, monoamine oxidase inhibitors and verapamil) or exposure to these drugs 30 days prior to placement on the study.
7. Concomitant use of vasoconstrictive nasal decongestants (e.g., oxymetazoline, phenylephrine, xylometazoline)
8. Numeric Rating Scale (NRS) pain score more than 0 at baseline
9. Any situation or condition which, in the investigator's opinion, puts the subject at significant risk, or could confound the study results.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2016-05-10 (Actual); Study Completion 2016-05-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain numeric rating scale | within 3 hours post administration of the drug
  The primary endpoint is the worst pain experienced at any time during the procedure.
  Pain will be assessed using the Numeric Rating Scale (NRS score 0 = no pain to 10 = worst possible pain).

SECONDARY OUTCOMES:
Oxyhemoglobin saturation | Every 5 minutes post administration of the drug until 3 hours
  Pulse oximetry will be recorded at baseline and every 5 minutes for 3 hours post drug-administration.

OTHER OUTCOMES:
Mean arterial blood pressure | every 15 minutes until 3 hours post drug-administration
  Will be recorded at baseline and every 15 minutes for 3 hours post drug-administration.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Reznichek, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Urology Clinic, Harbor-UCLA Medical Center, Torrance, California, United States

REFERENCES:
- [Background] Patel AR, Jones JS, Babineau D. Lidocaine 2% gel versus plain lubricating gel for pain reduction during flexible cystoscopy: a meta-analysis of prospective, randomized, controlled trials. J Urol. 2008 Mar;179(3):986-90. doi: 10.1016/j.juro.2007.10.065. Epub 2008 Jan 18. PMID 18206920
- [Background] Taghizadeh AK, El Madani A, Gard PR, Li CY, Thomas PJ, Denyer SP. When does it hurt? Pain during flexible cystoscopy in men. Urol Int. 2006;76(4):301-3. doi: 10.1159/000092051. PMID 16679829
- [Background] Calleary JG, Masood J, Van-Mallaerts R, Barua JM. Nitrous oxide inhalation to improve patient acceptance and reduce procedure related pain of flexible cystoscopy for men younger than 55 years. J Urol. 2007 Jul;178(1):184-8; discussion 188. doi: 10.1016/j.juro.2007.03.036. Epub 2007 May 17. PMID 17499771
- [Background] Song YS, Song ES, Kim KJ, Park YH, Ku JH. Midazolam anesthesia during rigid and flexible cystoscopy. Urol Res. 2007 Jun;35(3):139-42. doi: 10.1007/s00240-007-0091-7. Epub 2007 Apr 6. PMID 17415555
- [Background] Hruby G, Ames C, Chen C, Yan Y, Sagar J, Baron P, Landman J. Assessment of efficacy of transcutaneous electrical nerve stimulation for pain management during office-based flexible cystoscopy. Urology. 2006 May;67(5):914-7. doi: 10.1016/j.urology.2005.11.043. PMID 16698351
- [Background] Striebel HW, Koenigs D, Kramer J. Postoperative pain management by intranasal demand-adapted fentanyl titration. Anesthesiology. 1992 Aug;77(2):281-5. doi: 10.1097/00000542-199208000-00010. PMID 1642347
- [Background] Striebel HW, Pommerening J, Rieger A. Intranasal fentanyl titration for postoperative pain management in an unselected population. Anaesthesia. 1993 Sep;48(9):753-7. doi: 10.1111/j.1365-2044.1993.tb07583.x. PMID 8214490
- [Background] Striebel HW, Olmann T, Spies C, Brummer G. Patient-controlled intranasal analgesia (PCINA) for the management of postoperative pain: a pilot study. J Clin Anesth. 1996 Feb;8(1):4-8. doi: 10.1016/0952-8180(95)00167-0. PMID 8695078
- [Background] Striebel HW, Oelmann T, Spies C, Rieger A, Schwagmeier R. Patient-controlled intranasal analgesia: a method for noninvasive postoperative pain management. Anesth Analg. 1996 Sep;83(3):548-51. doi: 10.1097/00000539-199609000-00019. PMID 8780279
- [Background] Striebel HW, Kramer J, Luhmann I, Rohierse-Hohler I, Rieger A. [Pharmacokinetics of intranasal Fentanyl.]. Schmerz. 1993 Jun;7(2):122-5. doi: 10.1007/BF02527870. No abstract available. German. PMID 18415433
- [Background] Toussaint S, Maidl J, Schwagmeier R, Striebel HW. Patient-controlled intranasal analgesia: effective alternative to intravenous PCA for postoperative pain relief. Can J Anaesth. 2000 Apr;47(4):299-302. doi: 10.1007/BF03020941. PMID 10764171
- [Background] Saunders M, Adelgais K, Nelson D. Use of intranasal fentanyl for the relief of pediatric orthopedic trauma pain. Acad Emerg Med. 2010 Nov;17(11):1155-61. doi: 10.1111/j.1553-2712.2010.00905.x. PMID 21175512
- [Background] Borland M, Jacobs I, King B, O'Brien D. A randomized controlled trial comparing intranasal fentanyl to intravenous morphine for managing acute pain in children in the emergency department. Ann Emerg Med. 2007 Mar;49(3):335-40. doi: 10.1016/j.annemergmed.2006.06.016. Epub 2006 Oct 25. PMID 17067720
- [Background] Borland ML, Bergesio R, Pascoe EM, Turner S, Woodger S. Intranasal fentanyl is an equivalent analgesic to oral morphine in paediatric burns patients for dressing changes: a randomised double blind crossover study. Burns. 2005 Nov;31(7):831-7. doi: 10.1016/j.burns.2005.05.001. Epub 2005 Jul 6. PMID 16005154
- [Background] Foster D, Upton R, Christrup L, Popper L. Pharmacokinetics and pharmacodynamics of intranasal versus intravenous fentanyl in patients with pain after oral surgery. Ann Pharmacother. 2008 Oct;42(10):1380-7. doi: 10.1345/aph.1L168. Epub 2008 Aug 26. PMID 18728103
- [Background] Christrup LL, Foster D, Popper LD, Troen T, Upton R. Pharmacokinetics, efficacy, and tolerability of fentanyl following intranasal versus intravenous administration in adults undergoing third-molar extraction: a randomized, double-blind, double-dummy, two-way, crossover study. Clin Ther. 2008 Mar;30(3):469-81. doi: 10.1016/j.clinthera.2008.03.001. PMID 18405786
- [Background] Fuhr U. Drug interactions with grapefruit juice. Extent, probable mechanism and clinical relevance. Drug Saf. 1998 Apr;18(4):251-72. doi: 10.2165/00002018-199818040-00002. PMID 9565737
- [Background] Baele P, Kestens-Servaye Y, Goenen M. MAOI and cardiac surgery. Can J Anaesth. 1993 Jun;40(6):579-80. doi: 10.1007/BF03009749. No abstract available. PMID 8403128
- [Background] Gillman PK. Monoamine oxidase inhibitors, opioid analgesics and serotonin toxicity. Br J Anaesth. 2005 Oct;95(4):434-41. doi: 10.1093/bja/aei210. Epub 2005 Jul 28. PMID 16051647
- [Background] Noble WH, Baker A. MAO inhibitors and coronary artery surgery: a patient death. Can J Anaesth. 1992 Dec;39(10):1061-6. doi: 10.1007/BF03008376. PMID 1464133
- [Background] Dale O, Hjortkjaer R, Kharasch ED. Nasal administration of opioids for pain management in adults. Acta Anaesthesiol Scand. 2002 Aug;46(7):759-70. doi: 10.1034/j.1399-6576.2002.460702.x. PMID 12139528
- [Background] Fisher A, Watling M, Smith A, Knight A. Pharmacokinetics and relative bioavailability of fentanyl pectin nasal spray 100 - 800 microg in healthy volunteers. Int J Clin Pharmacol Ther. 2010 Dec;48(12):860-7. doi: 10.5414/cpp48860. PMID 21084042
- [Background] Hansen MS, Mathiesen O, Trautner S, Dahl JB. Intranasal fentanyl in the treatment of acute pain--a systematic review. Acta Anaesthesiol Scand. 2012 Apr;56(4):407-19. doi: 10.1111/j.1399-6576.2011.02613.x. Epub 2012 Jan 19. PMID 22260169
- [Background] Panagiotou I, Mystakidou K. Intranasal fentanyl: from pharmacokinetics and bioavailability to current treatment applications. Expert Rev Anticancer Ther. 2010 Jul;10(7):1009-21. doi: 10.1586/era.10.77. PMID 20645689
- [Background] Prommer E, Thompson L. Intranasal fentanyl for pain control: current status with a focus on patient considerations. Patient Prefer Adherence. 2011 Mar 18;5:157-64. doi: 10.2147/PPA.S7665. PMID 21573046
- [Background] Kress HG, Oronska A, Kaczmarek Z, Kaasa S, Colberg T, Nolte T. Efficacy and tolerability of intranasal fentanyl spray 50 to 200 microg for breakthrough pain in patients with cancer: a phase III, multinational, randomized, double-blind, placebo-controlled, crossover trial with a 10-month, open-label extension treatment period. Clin Ther. 2009 Jun;31(6):1177-91. doi: 10.1016/j.clinthera.2009.05.022. PMID 19695386
- [Background] Mercadante S, Radbruch L, Davies A, Poulain P, Sitte T, Perkins P, Colberg T, Camba MA. A comparison of intranasal fentanyl spray with oral transmucosal fentanyl citrate for the treatment of breakthrough cancer pain: an open-label, randomised, crossover trial. Curr Med Res Opin. 2009 Nov;25(11):2805-15. doi: 10.1185/03007990903336135. PMID 19792837
- [Background] Chung F. Discharge criteria--a new trend. Can J Anaesth. 1995 Nov;42(11):1056-8. doi: 10.1007/BF03011083. PMID 8590498
- [Background] Callahan CM, Unverzagt FW, Hui SL, Perkins AJ, Hendrie HC. Six-item screener to identify cognitive impairment among potential subjects for clinical research. Med Care. 2002 Sep;40(9):771-81. doi: 10.1097/00005650-200209000-00007. PMID 12218768